CLINICAL TRIAL: NCT06090552
Title: I CAN DO Surgical ACP (Improving Completion, Accuracy, and Dissemination of Surgical Advanced Care Planning) Trial
Brief Title: I CAN DO Surgical ACP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Irvine (Other); University of Minnesota (Other); National Institute on Aging (NIA) (NIH); Fairview University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P0562156; 1UG3AG081663-01 (NIH)
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Surgical Advanced Care Planning
MeSH Terms: interventions — College Fraternities and Sororities

STUDY DESIGN:
Intervention Model Description: 1:1:1 simple randomized block design stratified by enrollment site
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Letter, AD, PREPARE (Other): Letter about ACP, PREPARE advanced directive (AD), PREPARE website
  Interventions: Behavioral: Letter; Behavioral: AD; Behavioral: PREPARE website
- Letter, AD, PREPARE, reminders (Other): Letter, AD, PREPARE plus reminder messages
  Interventions: Behavioral: Letter; Behavioral: AD; Behavioral: PREPARE website; Behavioral: reminders
- Letter, AD, PREPARE, reminders, healthcare navigator (Other): Letter, AD, PREPARE website plus reminders plus a healthcare navigator on ACP documentation (clinically meaningful ACP, primary outcome)
  Interventions: Behavioral: Letter; Behavioral: AD; Behavioral: PREPARE website; Behavioral: reminders; Behavioral: healthcare navigator

INTERVENTIONS:
Behavioral: Letter — Letter about ACP
Behavioral: AD — PREPARE advanced directive (AD)
Behavioral: PREPARE website — PREPARE website
Behavioral: reminders — reminders to complete the advance directive
  Arms: Letter, AD, PREPARE, reminders; Letter, AD, PREPARE, reminders, healthcare navigator
Behavioral: healthcare navigator — healthcare navigators provide assistance to complete the advance directive
  Arms: Letter, AD, PREPARE, reminders, healthcare navigator

SUMMARY:
The goal of the Advanced Care Planning (ACP) study is to encourage patients aged 65 or older who are referred for elective surgery to have advanced care planning.

DETAILED DESCRIPTION:
ACP is also a critical way to support older adults in participating actively with clinicians in making real-time, complex medical decisions so that the medical care they receive is aligned with their goals. Our team has designed and tested a theory-based, interactive ACP patient-facing technology solution (PREPARE) based on the new ACP paradigm of preparing people for communication and medical decision-making. The study team hypothesizes that by including PREPARE into the EHR-centric pre-surgery workflow for older adults and including automated patient reminders, easy-to-read materials, and, in Arm 3, directed support from a healthcare navigator (HCN), they can empower patients and surgical teams to engage in ACP discussions. They also hypothesize that ACP documentation will increase more with increasing resource intensity (i.e., Arm 3 more than Arm 2 more than Arm 1).

Participants will be randomized to Arms: (1) Letter about ACP, PREPARE advanced directive (AD), PREPARE website; (2) Letter, advanced directive (AD), PREPARE plus reminder messages; (3) Letter, advanced directive (AD,) PREPARE plus reminders plus a healthcare navigator on ACP documentation (clinically meaningful ACP, primary outcome). All patients randomized to the intervention will be sent a patient-reported ACP engagement survey (secondary outcome).

ELIGIBILITY:
Inclusion Criteria:

- Older Adults (age 65+) referred for surgical evaluation

Exclusion Criteria:

1. ACP on file within 3 years prior to surgery (UCSF and UCI) and 5 years (UMN)
2. Was previously randomized into intervention for a prior surgery during the 18-month study period

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with clinically meaningful Advanced Care Planning | 6 months
  clinically meaningful ACP documentation (ACP-specific clinical notes, problem lists, Epic Smartforms or Smartphrases, advanced directives, Physician Orders for Life Sustaining Treatment, out of hospital do-not-resuscitate order, living wills, or CPT billing codes) available in the HCS EHR within 6 months of intervention.

SECONDARY OUTCOMES:
Patient Engagement Scores | 6 months
  Patient-centered outcomes will be derived from the validated 4-item ACP Engagement Survey.The survey will be administered 2 weeks after the pre-surgical clinic visit and a follow up survey will be sent 6 months later.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Wick, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, Irvine, Irvine, California
  - University of California, San Francisco, San Francisco, California
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
De-identified data sets are available at request at the conclusion of the study

REFERENCES:
- [Derived] Welton L, Colley A, Sudore RL, Melton GB, Botsford C, Oreper S, O'Brien SE, Koopmeiners JS, Gibbs L, Carmichael JC, Wick EC. I CAN DO Surgical ACP (Improving Completion, Accuracy and Dissemination of Surgical Advanced Care Planning): a protocol for a multisite, single-blinded, pragmatic randomised controlled trial to improve ACP completion in older adults in the presurgical setting. BMJ Open. 2025 Sep 23;15(9):e108850. doi: 10.1136/bmjopen-2025-108850. PMID 40987739